CLINICAL TRIAL: NCT06226792
Title: Muscle Architecture in Ankylosing Spondylitis and Its Relationship With Clinical Parameters
Brief Title: Muscle Architecture in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/340
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ankylosing Spondylitis; Muscle Weakness; Rheumatic Diseases
MeSH Terms: conditions — Spondylitis, Ankylosing; Muscle Weakness; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankylosing Spondylitis: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI), Bath Ankylosing Spondylitis Metrology Index (BASMI), Rivermead Mobility Index (RMI) will be evaluated.
  Vastus Lateralis, Tibialis Anterior, Lateral Gastrocnemius and Medial Gastrocnemius ultrasonography will be performed to evaluate muscle thickness, pennation angle and fascicle length.
  Isometric knee extension, isometric ankle dorsiflexion and isometric ankle plantar flexion strength will be evaluated with hand held dynamometer.
- Volunteers: Voluntary participants will be admitted to this group. Vastus Lateralis, Tibialis Anterior, Lateral Gastrocnemius and Medial Gastrocnemius ultrasonography will be performed to evaluate muscle thickness, pennation angle and fascicle length.
  Isometric knee extension, isometric ankle dorsiflexion and isometric ankle plantar flexion strength will be evaluated with hand held dynamometer.

SUMMARY:
The goal of this observational study is to determine whether there is a decrease in muscle mass and the relationship between lower extremity skeletal muscle mass, muscle strength and disease activity in Ankylosing spondylitis.

The main questions it aims to answer are:

* Is there a relationship between the muscle thickness and pennation angle of the quadriceps, Gastrocnemius medialis and lateralis, Vastus medialis and lateralis and tibialis anterior muscles with disease activity and muscle strength?
* Are there any differences in the results of morphological parameters of lower extremity muscles between Ankylosing spondylitis and voluntary participants? Researchers will compare voluntary participants to see if any difference in lower muscle morphological parameters.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) Ankylosing spondylitis (AS) is a systemic inflammatory rheumatic disease that can cause characteristic inflammatory low back pain and structural and functional disorders by affecting the axial and peripheral skeleton.

Functional impairment increases with age, disease duration, and severity of symptoms. It has been shown that there is a significant relationship between dysfunction and activity limitation in AS patients.

Recent studies have reported that both sarcopenia and decreased muscle strength occur in patients with chronic inflammatory diseases such as rheumatoid arthritis3. There are concerns that sarcopenia may affect exercise tolerance, activities of daily living, and ultimately have a negative impact on cardiovascular fitness and physical and emotional well-being. Given the risk of chronic inflammation and reduced physical activity, patients are also at risk of accelerated muscle wasting. In chronic diseases, loss of muscle mass, often referred to as cachexia, is a relevant systemic complication that leads to decreased muscle strength and endurance, reduced physical activity and fitness.

However, there is no study reporting variation in lower extremity information, muscle development, morphological effects measured by ultrasound, muscle strength and disease intensity in AS patients. Therefore, this study was conducted to determine whether there is a decrease in muscle according to the wide general spread in AS patients and to strengthen the detachable lower extremity structure with AS, muscle strength and possible presence. The relationship between strength, power and mobility of skeletal muscles was also evaluated. Although muscle loss was not morphologically evident in previous ultrasounds, it has not been investigated whether this leads to loss of muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥18 years old,
* Being diagnosed with AS according to The Assesment of Spondyloarthritis international society (ASAS) criteria
* Ability to giving consent
* Ability to live independently
* Ability to walk without assistive devices.

Exclusion Criteria:

* History of surgery on the spine or lower extremities,
* History of inflammatory rheumatic disease,
* Severe cardiovascular disease,
* Neuromuscular disease affecting muscle strength,
* Individuals following a regular exercise program,
* Secondary osteoarthritis.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients who applied to the Bezmialem Vakıf University, Physical Medicine and Rehabilitation Outpatient Clinic appropriate for eligibility criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 1 Day
  It evaluates disease-specific symptoms such as fatigue, spinal and peripheral joint pain, swelling and morning stiffness and is interpreted on a score ranging from 0 to 10. Each question is scored on a scale of 0 to 10. Aside from the last question, 0 indicates none and 10 indicate very severe. For the last question, 0 is 0 hours, 5 is one hour, and 10 is two or more hours.
  To calculate the BASDAI score, the formula is:
  BASDAI = ((Q1 + Q2 + Q3 + Q4) + ((Q5 + Q6) / 2)) / 5
Bath Ankylosing Spondylitis Functional Index (BASFI) | 1 Day
  It is an index that is fast and easy to apply, sensitive to changes and reliable, developed for determining and monitoring the functional status of patients with AS. It consists of 10 questions that evaluate patients' abilities to bend, reach, stand, change positions, climb stairs, and cope with activities of daily living. For each question, the final score is obtained by dividing the total score by 10 using the visual analogue scale (VAS) in the range of 0-10 cm. A higher score indicates a higher degree of functional limitations.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | 1 Day
  BASMI consists of five clinical measurements: cervical rotation, tragus wall distance, lumbar flexion, trunk lateral flexion, and intermalleolar distance. It was first developed as a two-point scale in 1994 and was later adapted to a 10-point score. The 10-point BASMI scale was used in our study.The higher the BASMI score the more severe the patient's limitation of movement due to their Ankylosing Spondylitis.
Rivermead Mobility Index | 1 Day
  It is a one-dimensional index that focuses on measuring mobility status and includes basic mobility activities. It includes a series of hierarchical activities, from turning over in bed to running, consisting of 14 questions and one observation that fit the Guttman Scale. RMI was mainly developed for the purpose of evaluating the results of physiotherapy interventions after head trauma or stroke, and it is reported that it can be used in hospitals, outpatient clinics or home environments without requiring expertise. Self-reporting is essential in answering questions. Only the 5th item is observed and evaluated by the interviewer. 1 point is given for each "yes" answer and a range of 0-15 points can be received. A score of 15 points indicates that there is no problem in mobility, and a score of 14 points and below indicates that there is a mobility problem.
Isometric Knee Extension Muscle Strength | 1 Day
  Isometric Knee Extension Muscle Strength will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Isometric Ankle Dorsiflexion Muscle Strength | 1 Day
  Isometric Ankle Dorsiflexion Muscle Strength will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Isometric Ankle Plantar Flexion Muscle Strength | 1 Day
  Isometric Ankle Plantar Flexion Muscle Strength will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Serkan Kılıçoğlu, Ass.Prof., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Glass NA, Torner JC, Frey Law LA, Wang K, Yang T, Nevitt MC, Felson DT, Lewis CE, Segal NA. The relationship between quadriceps muscle weakness and worsening of knee pain in the MOST cohort: a 5-year longitudinal study. Osteoarthritis Cartilage. 2013 Sep;21(9):1154-9. doi: 10.1016/j.joca.2013.05.016. PMID 23973125
- [Background] Walton JM, Roberts N, Whitehouse GH. Measurement of the quadriceps femoris muscle using magnetic resonance and ultrasound imaging. Br J Sports Med. 1997 Mar;31(1):59-64. doi: 10.1136/bjsm.31.1.59. PMID 9132215
- [Background] Blum D, Rodrigues R, Geremia JM, Brenol CV, Vaz MA, Xavier RM. Quadriceps muscle properties in rheumatoid arthritis: insights about muscle morphology, activation and functional capacity. Adv Rheumatol. 2020 May 19;60(1):28. doi: 10.1186/s42358-020-00132-w. PMID 32429993
- [Background] Aily JB, de Noronha M, de Almeida AC, Pedroso MG, Maciel JG, Mattiello-Sverzut AC, Mattiello SM. Evaluation of vastus lateralis architecture and strength of knee extensors in middle-aged and older individuals with knee osteoarthritis. Clin Rheumatol. 2019 Sep;38(9):2603-2611. doi: 10.1007/s10067-019-04539-9. Epub 2019 Apr 23. PMID 31016579
- [Background] Rastelli F, Capodaglio P, Orgiu S, Santovito C, Caramenti M, Cadioli M, Falini A, Rizzo G, Lafortuna CL. Effects of muscle composition and architecture on specific strength in obese older women. Exp Physiol. 2015 Oct;100(10):1159-67. doi: 10.1113/EP085273. Epub 2015 Sep 10. PMID 26279270
- [Background] van der Heijde D, Braun J, Deodhar A, Baraliakos X, Landewe R, Richards HB, Porter B, Readie A. Modified stoke ankylosing spondylitis spinal score as an outcome measure to assess the impact of treatment on structural progression in ankylosing spondylitis. Rheumatology (Oxford). 2019 Mar 1;58(3):388-400. doi: 10.1093/rheumatology/key128. PMID 29860356
- [Background] Wang CY, Olson SL, Protas EJ. Test-retest strength reliability: hand-held dynamometry in community-dwelling elderly fallers. Arch Phys Med Rehabil. 2002 Jun;83(6):811-5. doi: 10.1053/apmr.2002.32743. PMID 12048660
- [Background] Blazevich AJ, Cannavan D, Coleman DR, Horne S. Influence of concentric and eccentric resistance training on architectural adaptation in human quadriceps muscles. J Appl Physiol (1985). 2007 Nov;103(5):1565-75. doi: 10.1152/japplphysiol.00578.2007. Epub 2007 Aug 23. PMID 17717119